CLINICAL TRIAL: NCT03552770
Title: Single or Combined Protocols for the Treatment of Patients With Neovascular Age-related Macular Degeneration: Compliance, Risk/Benefit and Cost/Benefit Ratios
Brief Title: Single or Combined Protocols for NV-AMD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Collaborators: Regione Emilia-Romagna (Other)
Responsible Party: Principal Investigator, Francesco Parmeggiani, Medical Doctor - Associate Professor, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PRUA2-2013-00002008
Record Dates: First submitted 2018-05-28; First posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-06

CONDITIONS: Age-Related Macular Degeneration
Keywords: neovascular age-related macular degeneration; bevacizumab; pro-re-nata regimens; clinical governance
MeSH Terms: conditions — Macular Degeneration | interventions — Bevacizumab

STUDY DESIGN:
Intervention Model Description: The enrolled patients are randomized to the following therapeutic regimens: i. group A, a single intra-vitreous injection of bevacizumab pro-re-nata repeated after monthly periodic monitoring of the patient (IVIBx1 regimen); ii. group B, two combined intra-vitreous injections of bevacizumab, spaced 30 ± 10 days apart and pro-re-nata repeated after periodic monitoring of the patient (IVIBx2 regimen).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVIBx1 (Active Comparator): Patients treated with a single intra-vitreous injection of bevacizumab (1.25 mg in 0.05 ml of solution) pro-re-nata repeated after monthly periodic monitoring of each patient
  Interventions: Drug: Bevacizumab
- IVIBx2 (Active Comparator): Patients treated with two combined intra-vitreous injections of bevacizumab, (1.25 mg in 0.05 ml of solution) spaced 30 ± 10 days apart and pro-re-nata repeated after periodic monitoring of each patient
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — pro-re-nata repeated single or combined intra-vitreous injection of bevacizumab
  Other Names: intra-vitreous injection of bevacizumab

SUMMARY:
The present interventional study represents a Research Program for the Clinical Governance supported by supported by the Healthcare Fund of the Emilia-Romagna Region. It aims to evaluate, after 12 months of monitoring, clinical safety, therapeutic efficacy, number of intra-vitreous injections of bevacizumab (IVIB), compliance and quality of life correlated to the vision by comparing the data obtained in two groups of patients (group A and group B), affected by neovascular age-related macular degeneration (NV-AMD) never previously treated or already undergoing pro-re-nata (PRN) treatments with biological drugs inhibiting vascular endothelial growth factor (Vascular Endothelial Growth Factor, VEGF), i.e. anti-VEGF drugs. Participating patients are randomized to the following therapeutic regimens: i. group A, a single intra-vitreous injection of bevacizumab PRN repeated after monthly periodic monitoring of the patient (IVIBx1 regimen); ii. group B, two combined intra-vitreous injections of bevacizumab, spaced 30 ± 10 days apart and repeated as-needed after periodic monitoring of the patient (IVIBx2 regimen). Within the aforementioned regimens, the re-treatment (single or combined in patients undergoing IVIBx1 or IVIBx2, respectively) is performed when signs of persistent neovascular activity is present. The present trial consists of a randomized controlled open-label study with parallel arms to evaluate the non-inferiority of clinical safety and therapeutic efficacy of the IVIBx1 regimen compared to the IVIBx2 regimen (1: 1 allocation) administered in patients with NV-AMD. The number and type of tests, as well as the number of intra-vitreous injections of anti-VEGF drug performed in patients treated with the PRN regimens IVIBx1 or IVIBx2 do not differ from those performed during normal clinical practice at the Eye Clinic of the University Hospital of Ferrara. The intra-vitreous administration of bevacizumab is performed in accordance with the guidelines of the Italian Ophthalmology Society.

ELIGIBILITY:
Inclusion Criteria:

* age > 50 years
* ability to comply with study procedures
* active NV-AMD in either treatment-naïve or previously treated patients
* BCVA > 20/200 in the study eye

Exclusion Criteria:

* any other possible cause of choroidal neovascularization other than AMD
* ocular media opacities or other causes counteracting data collection
* presence or onset of contraindications to the use of bevacizumab

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2014-11-23 (Actual); Primary Completion 2016-11-24 (Actual); Study Completion 2016-12-29 (Actual)

PRIMARY OUTCOMES:
comparison of the mean modifications of the maximal visual acuity (BCVA, Best-Corrected Visual Acuity) between the IVIBx1 study group with respect to those registered in the IVIBx2 one | 12 months
  verify the "non-inferiority" of the therapeutic efficacy of the IVIBx2 regimen versus IVIBx1 regimen, considering the mean modification of the maximal visual acuity (BCVA, Best-Corrected Visual Acuity)
comparison of the number of intra-vitreous injections of bevacizumab (IVIB) between the IVIBx1 study group with respect to those performed in the IVIBx2 one | 12 months
  verify the "non-inferiority" of the therapeutic responsiveness of the IVIBx2 regimen versus IVIBx1 regimen, considering the number of intra-vitreous injections of bevacizumab (IVIB)
comparison of the number of non-severe adverse events (NSAE) between the IVIBx1 study group with respect to those registered in the IVIBx2 one | 12 months
  verify the "non-inferiority" of the tolerability of the IVIBx2 regimen versus IVIBx1 regimen, considering the number of non-severe adverse events (NSAE)
comparison of the number of severe adverse events (SAE) between the IVIBx1 study group with respect to those registered in the IVIBx2 one | 12 months
  verify the "non-inferiority" of the safety of the IVIBx2 regimen versus IVIBx1 regimen, considering the number of severe adverse events (SAE)

SECONDARY OUTCOMES:
comparison of the number of unjustified absences of patients at the diagnostic checks and/or therapeutic procedures between the IVIBx1 study group with respect to those registered in the IVIBx2 one | 12 months
  verify the "non-inferiority" of the objective patient's compliance during the IVIBx2 regimen versus IVIBx1 regimen, considering the number of unjustified absences of patients at the diagnostic checks and/or therapeutic procedures foreseen by the study
comparison of the mean modifications of the score of the National Eye Institute Visual Functioning Questionnaire (NEI-VFQ) between the IVIBx1 study group with respect to those registered in the IVIBx2 one | 12 months
  verify the "non-inferiority" of the vision-related quality of life during the IVIBx2 regimen versus IVIBx1 regimen, considering the mean modification of the score of the National Eye Institute Visual Functioning Questionnaire (NEI-VFQ)
comparison of the mean modification of the score of a specific questionnaire about patient's satisfaction for the received care between the IVIBx1 study group with respect to those registered in the IVIBx2 one | 12 months
  verify the "non-inferiority" of the subjective patient's compliance during the IVIBx2 regimen versus IVIBx1 regimen, considering the mean modification of the score of a specific questionnaire about the assessment of patient satisfaction with respect to the received healthcare

IPD SHARING:
Plan to Share IPD: No